CLINICAL TRIAL: NCT00050505
Title: A Multicenter, Double Blind, Randomized Dose-response Study of Dryvax Vaccine Against Smallpox in Previously Vaccinated Adults
Brief Title: Expanded Dryvax Dilution Study in Previously Vaccinated Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 02-007
Record Dates: First submitted 2002-12-10; First posted 2002-12-11 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2009-07

CONDITIONS: Smallpox
Keywords: smallpox, Dryvax, vaccine, dilution
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Cohort C (Experimental): N=100 to 110 subjects receives 1:10 diluted dose of Dryvax vaccine on Day 0 and 1:5 revaccination dose on Day 56
  Interventions: Biological: Live vaccinia virus vaccine
- Cohort B (Experimental): N=571 to 581 subjects receives 1:5 diluted dose of Dryvax vaccine on Day 0 and 1:5 revaccination dose on Day 56
  Interventions: Biological: Live vaccinia virus vaccine
- Cohort A (Experimental): N=226 to 236 subjects receives undiluted dose Dryvax vaccine on Day 0 and 1:5 revaccination dose on Day 56
  Interventions: Biological: Live vaccinia virus vaccine

INTERVENTIONS:
Biological: Live vaccinia virus vaccine — Dryvax undiluted. Cohort A receives undiluted dose of Dryvax vaccine
  Arms: Cohort A
Biological: Live vaccinia virus vaccine — Dryvax with diluent (50% glycerin and 0.25% phenol in sterile water). Cohort A-C receives diluted dose of Dryvax vaccine.

SUMMARY:
The purpose of this study is to determine the safety and effect of diluting smallpox vaccine, making a larger number of doses in case smallpox is released into the environment. A total of up to 927 healthy adults between the ages of 32 and 70 years who were already vaccinated against smallpox (but not since 1989) will volunteer for this study for up to 34 weeks and receive different strengths of vaccine. Some subjects may participate for longer if they choose to be revaccinated because the first vaccination does not take. The vaccine will be given by making small cuts in the skin and putting the vaccine into these cuts. After the screening visit, volunteers will be followed through study visits and follow up phone calls. Blood will be collected during some study visits to look at the immune system (body system that fights infection) response.

DETAILED DESCRIPTION:
The purposes of this multi-center, double blind randomized dose response study are: to evaluate the safety of undiluted Dryvax and Dryvax diluted at 1:5 and 1:10 in adults between the ages of 32 and 70 years who were previously vaccinated but not since 1989 and to define, with very high precision (+/-3%), the proportion of individuals who respond with a "take" 6 to 11 days after vaccination with undiluted Dryvax vaccine and Dryvax diluted at 1:5. A "take" is defined as the formation of a lesion at the site of vaccination that is consistent with the description of a successful vaccination described in the IB Secondary study objectives include defining with good precision (+/- 10%), the proportion of individuals who respond with a "take" 6 to 11 days after vaccination with a 1:10 dilution of Dryvax vaccine and exploring correlations between "takes"/ no-"take" and immune responses in all vaccine groups (antibody responses in all volunteers; and assays of cell-mediated immunity in a convenience sample consisting of 15 volunteers enrolled at each site (total N = 105) randomly distributed across the vaccine groups). Immunogenicity assays will include neutralizing antibody to vaccinia, vaccinia binding antibody, ELISPOT for gamma interferon [Assays of cell-mediated immunity will be performed only on a convenience sample consisting of 15 volunteers enrolled at each site (total N = 105)] and intracellular cytokine production. Primary safety endpoints include safety data regarding the three doses of vaccine in previously vaccinated subjects as assessed by adverse events reported by the subjects and/or investigators and changes observed during the scheduled clinic visits. Specific attention will be paid to the following: local reactogenicity at the site of injection: pain, tenderness, erythema, induration, regional lymphadenopathy, limitation of limb movement; systemic symptoms: fever, myalgia, fatigue, and headache; anaphylaxis, and hypersensitivity reactions; other reactions: dermatologic, neurologic, gastrointestinal (nausea/vomiting, diarrhea). The primary efficacy endpoint for this trial will be the proportion of vaccinees demonstrating a "take" 6 to 11 days after the first vaccination at each of the dose levels (undiluted and 1:5 and 1:10). Secondary endpoints are: immune responses as assessed by vaccinia neutralizing antibody measured on all subjects and binding antibody to vaccinia on all subjects and the size of the lesions observed in all subjects compared across the dilution groups. Tertiary endpoints of 15 volunteers at each site randomly distributed across the vaccine groups are cellular immune responses as assessed by: ELISPOT for gamma interferon in response to vaccinia antigens and intracellular cytokine production.

ELIGIBILITY:
Inclusion Criteria:

1. Age 32 to 70 years.
2. Typical vaccinia scar or validated documentation (e.g., military record, international travel certificate) of a smallpox vaccination, but not since 1989.
3. Willing to sign informed consent.
4. Availability for follow-up for the planned duration of the study (at least 26 weeks after vaccination).
5. Acceptable medical history by screening evaluation and brief clinical assessment.
6. Negative urine or serum pregnancy test for women of childbearing potential.
7. If the subject is female and of childbearing potential, she must use an acceptable contraception and not become pregnant within 56 days post vaccination. (Acceptable contraception includes implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).
8. Negative ELISA for HIV or indeterminant Western blot or other assay confirming that the serostatus does not reflect HIV infection
9. ALT < 1.5 times institutional upper limit of normal.
10. Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
11. Negative urine glucose by dipstick.
12. Adequate renal function defined as a serum creatinine less than or equal to 1.5 mg/dL; urine protein < 100 mg/dL or trace or negative proteinuria by dipstick; and a calculated creatinine clearance > 55 mL/min based on the formulas in the manual of procedures.
13. Hematocrit > 34% for females, > 38% for males; platelets > 150,000/mm3; and WBC > 2,500/mm3 and < 11,000/mm3.

Exclusion Criteria:

1. Smallpox vaccination in 1990 or more recently.
2. History of immunodeficiency.
3. Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
4. Malignancy, other than squamous cell or basal cell skin cancer.
5. Active autoimmune disease.
6. Use of immunosuppressive medication.
7. Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol.
8. History of "illegal" injection drug use.
9. Inactivated vaccine 14 days prior to vaccination
10. Live attenuated vaccines within 60 days of study.
11. Use of investigational agents within 30 days prior to study.
12. Receipt of blood products or immunoglobulin in the past 6 months.
13. Acute febrile illness on the day of vaccination.
14. Pregnant or lactating women.
15. Eczema of any degree or history of eczema.
16. History of chronic exfoliative skin disorders/conditions.
17. Any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2 x 2 cm.
18. Household contacts/sexual contacts with, or frequent and/or prolonged exposure to, any of the following:

    * Pregnant women
    * Children < 12 months of age
    * People with or history of eczema
    * People with chronic exfoliative skin disorders/conditions or any acute skin disorders of large magnitude. e.g., laceration requiring sutures, burn greater than 2 x 2 cm
    * People with immunodeficiency disease or use of immunosuppressive medications
19. Any condition that, in the opinion of the investigator, might interfere with study objectives.
20. Known allergies to any component of the vaccine (e.g., polymyxin B sulfate, dihyrostreptomycin sulfate, chlortetracycline hydrochloride, neomycin sulfate).
21. Known allergies to any known component of the diluent (i.e., glycerin and phenol).
22. Known allergies to any known component of VIG, i.e., thimerosal or previous allergic reaction to immunoglobulins.
23. Known allergies to cidofovir or probenecid.

Ages: 32 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2002-10; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Proportion of vaccinees demonstrating a "take" 6 to 11 days after the first vaccination at each of the dose levels (undiluted and 1:5 and 1:10). | 6 to 11 days after the first vaccination at each of the dose levels (undiluted and 1:5 and 1:10).

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - Stanford University, Stanford, California
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Duke Health Center, Durham, North Carolina